CLINICAL TRIAL: NCT06669325
Title: Role of Apfel's Score in Predicting Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: National Medical College Birgunj (Other)
Responsible Party: Principal Investigator, Rajendra Dhakal, Clinical Professor, National Medical College Birgunj
Other Study IDs: PG-NMC/541/078-079
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: APFEL RİSK SCORE; Post Operative Nausea and Vomiting (PONV)
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to assess the role of Apfel's score in predicting postoperative nausea and vomiting (PONV) after laparoscopic cholecystectomy in patients with symptomatic cholelithiasis. The main questions it aims to answer are:

1. Does Apfel's score accurately predict the occurrence of PONV after laparoscopic cholecystectomy?
2. Which components of Apfel's score are most strongly associated with PONV?

Participants will undergo laparoscopic cholecystectomy under general anesthesia. Researchers will calculate each participant's Apfel score preoperatively, and postoperative outcomes, such as nausea and vomiting, will be monitored for 24 to 48 hours. Researchers will compare PONV incidence among patients with varying Apfel scores to determine if higher scores correlate with a higher risk of PONV.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 90 years.
* Patient scheduled for elective laparoscopic cholecystectomy for symptomatic cholelithiasis.
* Patients who provided written informed consent to participate in the study.

Exclusion Criteria:

* Patients receiving prophylactic antiemetic medications prior to surgery.
* Patients on opioid analgesics for reasons other than the surgical procedure.
* Pregnant women.
* Patients whose laparoscopic cholecystectomy was converted to open cholecystectomy during the operation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients who are undergoing elective laparoscopic cholecystectomy for symptomatic cholelithiasis. These patients are treated at the Department of General Surgery at National Medical College Teaching Hospital, Birgunj, Nepal.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Nausea and Vomiting (PONV) | Assessed for 24 hours post-surgery.
  The number of patients who experience nausea and/or vomiting within 24 hours after laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
Relationship Between Apfel's Score and PONV Incidence | Assessed for 24 hours post-surgery.
  Evaluating the correlation between the Apfel's score (0-4) and the likelihood of PONV in patients after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical College and Teaching Hospital, Birgunj, Birgunj, Madesh, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
The investigators may share de-identified Individual Participant Data (IPD) with other researchers upon reasonable request. Access to the data will be granted after approval by the Institutional Review Committee, and a data-sharing agreement will be required to ensure participant confidentiality and compliance with ethical standards.